CLINICAL TRIAL: NCT00715208
Title: A Two-Arm, Non-Randomized, Multicenter, Phase 2 Study of VELCADE (Bortezomib) in Combination With Rituximab, Cyclophosphamide, and Prednisone With or Without Doxorubicin Followed by Rituximab Maintenance in Patients With Relapsed Follicular Lymphoma.
Brief Title: Phase 2 Study of VELCADE (Bortezomib) in Patients With Relapsed Follicular Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C05012
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Results first posted 2013-04-29 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Relapsed Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Bortezomib; Prednisone

ARMS (2):
- VELCADE R-CAP (Experimental): VELCADE will be administered as a 3- to 5-second intravenous bolus injection, rituximab 375 mg/m2 Intravenous on Day 1, cyclophosphamide 750 mg/m2 intravenous on Day 1, doxorubicin 50 mg/m2 intravenous on Day 1, VELCADE 1.6 mg/m2 intravenous on Days 1 and 8, prednisone 100 mg orally on Days 1 to 5 of a 21-day (3-week) cycle for 6 cycles.
  Interventions: Drug: rituximab; Drug: cyclophosphamide; Drug: doxorubicin; Drug: VELCADE; Drug: prednisone
- VELCADE R-CP (Experimental): VELCADE will be administered as a 3- to 5-second intravenous bolus injection, rituximab 375 mg/m2 intravenous on Day 1, cyclophosphamide 1000 mg/m2 intravenous on Day 1, VELCADE 1.6 mg/m2 intravenous on Days 1 and 8, prednisone 100 mg orally on Days 1 to 5 of a 21-day (3-week) cycle for 6 cycles.
  Interventions: Drug: rituximab; Drug: cyclophosphamide; Drug: VELCADE; Drug: prednisone

INTERVENTIONS:
Drug: rituximab
Drug: cyclophosphamide
Drug: doxorubicin
  Arms: VELCADE R-CAP
Drug: VELCADE
Drug: prednisone

SUMMARY:
This is a phase 2, two-arm, non-randomized, open-label, multicenter study evaluating the safety and efficacy of 2 VELCADE-containing regimens. Patients will be treated with either a combination of VELCADE, rituximab, cyclophosphamide, doxorubicin, and prednisone (VELCADE-R-CAP) or a combination of VELCADE, rituximab, cyclophosphamide, and prednisone (VELCADE-R-CP) based on investigator preference. Following completion of the treatment period, patients will receive maintenance therapy with rituximab up to a maximum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient 18 years of age or older
* Pathological diagnosis of follicular lymphoma (any grade) or marginal zone lymphoma. Patients with transformed follicular lymphoma are eligible, provided there has previously been pathologic documentation of follicular lymphoma.
* Documented relapse or progression following prior antineoplastic therapy
* At least 1 measurable tumor mass that is greater than 1.5 cm in the long axis and greater than 1.0 cm in the short axis that has not been previously irradiated, or has grown since previous irradiation
* No clinically significant evidence of active central nervous system lymphoma
* Karnofsky performance status (KPS) ≥50 (equivalent to Eastern Cooperative Group Oncology Group [ECOG] status ≤2)

Exclusion Criteria:

* Diagnosed or treated for a malignancy other than Non-Hodgkin's Lymphoma (NHL) within 2 years of first dose, or who were previously diagnosed with a malignancy other than NHL and have any radiographic or biochemical marker evidence of malignancy. Patients with prostate cancer who were treated with definitive radiotherapy who have a serum prostate-specific antigen <1 ng/mL are not excluded. Patients are not excluded if they have had basal cell or squamous cell carcinoma of the skin that was completely resected, or any in situ malignancy that was adequately treated.
* Received any of the following treatments or procedures outside of the specified timeframes:

  * Prior treatment with VELCADE
  * Prior treatment with a cumulative dose of doxorubicin of more than 100 mg/m2, if assigned to Arm A (VELCADE-R-CAP)
  * Antineoplastic (including unconjugated therapeutic antibodies and toxin immunoconjugates), experimental, or radiation therapy within 3 weeks before Day 1 of Cycle 1
  * Nitrosoureas within 6 weeks before Day 1 of Cycle 1
  * Radioimmunoconjugates within 10 weeks before Day 1 of Cycle 1
  * Autologous stem cell transplant within 3 months before Day 1 of Cycle 1, or prior allogeneic stem cell transplant at any time
  * Major surgery within 2 weeks before Day 1 of Cycle 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-09; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (43):
- United States (42):
  - Northwest Alabama Center, PC, Muscle Shoals, Alabama
  - Providence Saint Joseph Medical Center, Burbank, California
  - Pacific Coast Hematology Oncology Medical Group, Fountain Valley, California
  - Loma Linda U Cancer Center, Loma Linda, California
  - Desert Hematology Medical Group, Inc., Rancho Mirage, California
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Ocala Cancer Institute, Ocala, Florida
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - Southern Illinois Hematology Oncology, Centralia, Illinois
  - Alexian Brothers Hospital Network, Elk Grove Village, Illinois
  - Clintell, Inc., Skokie, Illinois
  - Cancer Care Center, Inc., New Albany, Indiana
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Hutchinson Clinic, Hutchinson, Kansas
  - Purchase Cancer Group, Paducah, Kentucky
  - Medical Oncology, LLC, Baton Rouge, Louisiana
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - Kalamazoo Hematology and Oncology, Kalamazoo, Michigan
  - Jackson Oncology Associates, PLLC, Jackson, Mississippi
  - St. Louis Cancer Care, LLP, Chesterfield, Missouri
  - Nebraska Hematology-Oncology, PC, Lincoln, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - San Juan Oncology Associates, Farmington, New Mexico
  - NYU Clinical Cancer Center, New York, New York
  - Interlakes Foundation, Rochester, New York
  - New York Medical College, Valhalla, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Oklahoma Oncology and Hematology, PC, Oklahoma City, Oklahoma
  - Oklahoma Oncology and Hematology, PC, Tulsa, Oklahoma
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - Landmark Medical Center, Woonsocket, Rhode Island
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - HOPE Oncology, Richardson, Texas
  - Northern Utah Associates, Ogden, Utah
  - Marshall University, Huntington, West Virginia
  - West Virginia University Health Science Center, Morgantown, West Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
- Auxilio Cancer Center, Hato Rey, Puerto Rico

REFERENCES:
- [Derived] Craig M, Hanna WT, Cabanillas F, Chen CS, Esseltine DL, Neuwirth R, O'Connor OA. Phase II study of bortezomib in combination with rituximab, cyclophosphamide and prednisone with or without doxorubicin followed by rituximab maintenance in patients with relapsed or refractory follicular lymphoma. Br J Haematol. 2014 Sep;166(6):920-8. doi: 10.1111/bjh.12991. Epub 2014 Jul 9. PMID 25039282

RESULTS

PARTICIPANT FLOW:
Groups:
- VELCADE R-CAP: VELCADE, rituximab, cyclophosphamide, prednisone, and Doxorubicin
- VELCADE R-CP: VELCADE, rituximab, cyclophosphamide, and prednisone
Period: Overall Study
Arm/Group | VELCADE R-CAP | VELCADE R-CP
Started | 7 | 48
Completed | 6 | 39
Not Completed | 1 | 9
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 6
Not completed — Lack of Efficacy | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VELCADE R-CAP | VELCADE R-CP | Total
Number analyzed (Participants) | 7 | 48 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 27 | 34
  >=65 years | 0 | 21 | 21
Age Continuous [Mean (Standard Deviation); unit: years] | 62.9 (8.30) | 62.3 (11.39) | 62.3 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 24 | 29
  Male | 2 | 24 | 26
Region of Enrollment [Number; unit: participants]
  United States | 7 | 48 | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Complete Response (CR)
Description: Disappearance of all evidence of disease assessed by computed tomography (CT) and PET (position-emission tomography) according to the revised International Working Group (IWG) Criteria.
Time Frame: 30 weeks
Population: Response evaluable: measurable disease at baseline, completed first scheduled response evaluation, or do not complete first scheduled response evaluation due to progressive disease (PD) or death.
Measure: Number; unit: participants
Arm/Group | VELCADE R-CAP | VELCADE R-CP
Number analyzed (Participants) | 6 | 48
participants | 1 [0 to 36] | 13

2. Secondary Outcome: Number of Participants With Overall Response (OR)
Description: OR = Complete Response (CR) + Partial Response (PR)according to the revised International Working Group (IWG) Criteria.
  CR is the disappearance of all evidence of disease assessed by CT and PET. PR is the regression of measurable disease and no new sites assessed by CT and PET.
Time Frame: 30 weeks
Population: Response evaluable: measurable disease at baseline, completed first scheduled response evaluation, or do not complete first scheduled response evaluation due to PD or death.
Measure: Number; unit: participants
Arm/Group | VELCADE R-CAP | VELCADE R-CP
Number analyzed (Participants) | 6 | 48
participants | 6 | 37

3. Secondary Outcome: Percentage of Participants With Progression-free Survival (PFS) at 1 Year
Description: PFS was defined as the time from the first dose to the date of progressive disease (PD)/relapse or death, whichever comes first. For a participant who had not progressed/relapsed or died, PFS was censored at the last response assessment that was stable disease (failure to attain complete response/partial response or PD or better).
Time Frame: Assessed at at the end of Cycle 2, at end of treatment visit, and every 12± 1 weeks for the first year (4 visits) until PD
Population: Safety population: Treated
Measure: Number; unit: percentage of participants
Arm/Group | VELCADE R-CAP | VELCADE R-CP
Number analyzed (Participants) | 7 | 48
percentage of participants | 67 [lower limit 9.4] | 63 [lower limit 11.2]

4. Secondary Outcome: Duration of Response
Description: Time (in months) from the first documentation of a response (CR or partial response [PR]) to the date of first documentation of progressive disease or relapse from complete response.
  CR is defined as disappearance of all evidence of disease assessed by CT or PET; PR is defined as regression of measurable disease and no new sites assessed by CT or PET according to the revised International Working Group (IWG) Criteria.
Time Frame: 2 years
Population: Responders: CR + PR (Not done for VELCADE R-CAP, only 5 responders)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | VELCADE R-CAP | VELCADE R-CP
Number analyzed (Participants) | 0 | 37
Months |  | 21.9 [9.4 to NA] — The upper endpoint is not estimable (NE). For subjects who had not progressed, duration of response was censored at the last response assessment that was stable disease (SD) or better.

5. Secondary Outcome: Number of Patients Who Experienced at Least One Serious Adverse Event
Time Frame: From completion of informed consent through 30 days after the last dose of study drug
Population: Safety Population: Treated patients
Measure: Number; unit: participants
Arm/Group | VELCADE R-CAP | VELCADE R-CP
Number analyzed (Participants) | 7 | 48
participants | 2 | 12

ADVERSE EVENTS:
Arm/Group | VELCADE R-CAP | VELCADE R-CP
Serious Adverse Events (participants affected / at risk) | 2/7 | 12/48
Other Adverse Events (participants affected / at risk) | 7/7 | 47/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VELCADE R-CAP (N=7) | VELCADE R-CP (N=48)
Bronchitis NOS (Infections and infestations) | 0 | 1
Bronchitis acute NOS (Infections and infestations) | 0 | 1
Pneumonia NOS (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0
Respiratory tract infection NOS (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Viral infection NOS (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 1 | 3
Fatigue (General disorders) | 0 | 1
Weakness (General disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2
Leukopenia NOS (Blood and lymphatic system disorders) | 1 | 0
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (excl neonatal) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Abdominal pain NOS (Gastrointestinal disorders) | 0 | 1
Blood culture positive (Investigations) | 0 | 2
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Headache NOS (Nervous system disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Hypertension aggravated (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VELCADE R-CAP (N=7) | VELCADE R-CP (N=48)
Diarrhoea (Gastrointestinal disorders) | 2 | 24
Nausea (Gastrointestinal disorders) | 3 | 21
Vomiting NOS (Gastrointestinal disorders) | 0 | 12
Constipation (Gastrointestinal disorders) | 3 | 10
Stomatitis (Gastrointestinal disorders) | 3 | 2
Pharyngolaryngeal pain (Gastrointestinal disorders) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 8
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3
Skin lesion NOS (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Rigors (General disorders) | 4 | 6
Oedema lower limb (General disorders) | 2 | 5
Fatigue aggravated (General disorders) | 1 | 5
Infusion associated symptoms (General disorders) | 0 | 3
Fall (General disorders) | 2 | 0
Chest pain (General disorders) | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 2 | 6
Dehydration (Metabolism and nutrition disorders) | 3 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 2
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 6
Lymphopenia (Blood and lymphatic system disorders) | 2 | 6
Peripheral neuropathy NOS (Nervous system disorders) | 2 | 10
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3
Peripheral neuropathy aggravated (Nervous system disorders) | 1 | 0
Dizziness (excl vertigo) (Nervous system disorders) | 2 | 7
Dysgeusia (Nervous system disorders) | 4 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Restless leg syndrome (Nervous system disorders) | 1 | 0
Upper respiratory tract infection NOS (Infections and infestations) | 0 | 8
Herpes zoster (Infections and infestations) | 1 | 3
Urinary tract infection NOS (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Rhinitis NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle cramps (Musculoskeletal and connective tissue disorders) | 2 | 1
Peripheral swelling (Musculoskeletal and connective tissue disorders) | 0 | 3
White blood cell count decreased (Investigations) | 1 | 4
Lymphocyte count decreased (Investigations) | 0 | 4
Neutrophil count decreased (Investigations) | 0 | 4
Haemoglobin decreased (Investigations) | 0 | 6
Blood uric acid increased (Investigations) | 0 | 4
Platelet count decreased (Investigations) | 0 | 4
Blood glucose increased (Investigations) | 0 | 3
Blood urea increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 7
Confusion (Psychiatric disorders) | 1 | 0
Hypotension NOS (Vascular disorders) | 2 | 2
Flushing (Vascular disorders) | 0 | 3
Lacrimation increased (Eye disorders) | 0 | 4
Eye irritation (Eye disorders) | 0 | 4
Tachycardia NOS (Cardiac disorders) | 1 | 1
Sinus Tachycardia (Cardiac disorders) | 1 | 2
Ventricular hypokinesia (Cardiac disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Hypoproteinaemia (Hepatobiliary disorders) | 1 | 1
Hypersensitivity NOS (Immune system disorders) | 1 | 0
Breast discomfort (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No